CLINICAL TRIAL: NCT01179412
Title: Treatment of Epidemic Keratoconjunctivitis With 2% Povidone-iodine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Adisak Trinavara t/ Associate Professor, Department of Ophthalmology, Siriraj Hospital Mahidol University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EKC2004
Record Dates: First submitted 2010-07-18; First posted 2010-08-11 (Estimated); Last update posted 2010-08-11 (Estimated); Status verified 2010-08

CONDITIONS: Viral Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Viral | interventions — Povidone-Iodine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 2% povidone-iodine (Experimental)
  Interventions: Drug: 2% povidone-iodine

INTERVENTIONS:
Drug: 2% povidone-iodine — apply 4 times a day for one week
  Other Names: PVP-I
Drug: 2% povidone-iodine — apply 2% povidone-iodine 4 times per day for one week
  Other Names: PVP-I

SUMMARY:
The purpose of this study is to determine the outcomes of treating epidemic keratoconjunctivitis with 2% povidone-iodine.

DETAILED DESCRIPTION:
The study design was a prospective interventional case series. Our institutional ethical committee approved the study protocol in April 2004. We performed this study between July 2004 and December 2009. During this period, there were 2 episodes of EKC epidemic. The first episode was in 2006 and the second in 2009.

ELIGIBILITY:
Inclusion Criteria:

* patients who were diagnosed with EKC at the outpatient ophthalmic unit

Exclusion Criteria:

* children younger than six years
* women being pregnant or during lactation
* history of allergy to povidone-iodine
* prior ocular surgery
* contact lens usage and chronic eye diseases with current eye medications.

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2004-07; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
the recovery rate within one week of treatment | 1 week

SECONDARY OUTCOMES:
drug tolerability | 1 week
  proportion of patient who can continue topical application of povidone-iodine for a week or until EKC subsides

CONTACTS AND LOCATIONS:
Overall Officials: Adisak Trinavarat, MD, Principal Investigator — Siriraj Hospital
Locations (1):
- Department of Ophthalmology, Siriraj Hospital Mahidol University, Bangkoknoi, Bangkok, Thailand